CLINICAL TRIAL: NCT00331357
Title: Cohort of Children With Acute Immune or Idiopathic Thrombocytopenic Purpura (ITP) : a Prospective Study in Pays De La Loire
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Ministry of Health, France (Other Government)
Other Study IDs: PHRC-05-06; CCPPRB : 2006/04; DGS : 2006/0212
Record Dates: First submitted 2006-05-29; First posted 2006-05-31 (Estimated); Last update posted 2006-05-31 (Estimated); Status verified 2006-05

CONDITIONS: Acute Idiopathic Thrombocytopenic Purpura
Keywords: acute idiopathic thrombocytopenic purpura; paediatric; quality of life

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The objective of this study is to describe a paediatric population presenting an acute idiopathic thrombocytopenic purpura (ITP) and their evolution during their therapy in the region Pays de la Loire. The study will particularly evaluate the quality of life of these patients and their parents.

The secondary objectives are to identify the predictive factors of the complications, the repetitions and the chronicity of the ITP, to estimate the principal parameters of the economic cost of therapy of the children suffering from ITP according to the protocol of therapy, set up in the region Pays de la Loire and the constitution of a blood sample collection which allow a better understanding of the physiopathology of this disease.

It is about a prospective, multicentric clinical epidemiologic study of a paediatric cohort. Patients: 100 children from 0 to 17,99 years suffering from a first discovered ITP. The patients are not included if they present a serious, intercurrent, stabilized chronic pathology or not likely to modify the quality of life of the child and if they present a pathology other than the thrombopenia bringing into play the vital prognosis within a time lower than one year. These patients will be followed for 6 months according to the diagnosis of their ITP.

During the 6 months follow-up of each patient, the study will not carry out more consultations, nor more blood tests than the usual follow-up of a child suffering from ITP. On the other hand, in addition to the J0 questionnaire, it will be requested to the patient and to his family to fill in the questionnaires of quality of life and way of life during the consultations of J8, 1 month, 3 months and 6 months. A check-up of autoimmunity at 6 months will be carried out if the thrombopenia persists (this check-up is usual and not-specific to the study). At the time of the blood test for the control of the platelets at J0 and 6 months, an additional blood sample will be carried out: 5 ml are taken for the children of an age ≤ at 2 years, 10 ml from 2 to 4 years and 15 ml of blood for the children of an age > at 4 years. These blood samples are intended for the constitution of a blood sample collection.

The protocol of therapy of the children suffering from ITP is homogeneous in all centers, this protocol being a consensus established by the network of Oncopaediatrics of the Pays de la Loire. The instituted treatment will be in function of the gravity of the ITP expressed in 4 stages:

Stage I: Platelets > 20 gigas/L and absence of clinical signs. Stage II: Platelets > 10 gigas/L and hemorrhagic signs: haematomas, petechias or occasional epistaxis without repercussion on the daily life.

Stage III: moderate. Platelets > 10.000/mm3 and epistaxis with gauze pluggings or mucous lesions.

Stage IV: severe. Platelets ≤ 10.000/mm3 or fall of 2 grs/dl of haemoglobin with bleedings: epistaxis, melaena or haemorrhages requiring a blood transfusion or an hospitalization and important changes in the activities of the daily life.

Stages I and II do not receive any treatment and benefit from a simple monitoring.

Stages III benefit from either a corticosteroid treatment (Méthylprednisolone or Prednisone) at the dose of 4 mg/kg and per day in 2 intervals during 4 days (maximal dose of 100 mg/day) or a monitoring according to the appreciation of the clinician.

Stages IV profit in first intention from a treatment by Méthylprednisolone or Prednisone at the dose of 4 mg/kg and per day in 2 intervals during 4 days (maximal dose of 100 mg/jour).

The therapeutic attitude and the stadification belong to a regional consensus, established before the study, but each one can decide to apply a treatment according to the gravity of the clinical state of the child.

ELIGIBILITY:
Inclusion Criteria:

* children 0 to 17,99 years
* suffering from a first discovered ITP

Exclusion Criteria:

* serious, intercurrent, stabilized chronic pathology or not likely to modify the quality of life of the child
* pathology other than the thrombopenia bringing into play the vital prognosis within a time lower than one year

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100
Dates: Start 2006-06; Study Completion 2008-12

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle PELLIER, MD, Study Director — UH of Angers
Locations (7):
- France (7):
  - UH of Angers, Angers
  - Hospital of Cholet, Cholet
  - Hospital of La Roche Sur Yon, La Roche-sur-Yon
  - Hospital of Laval, Laval
  - Hospital of Le Mans, Le Mans
  - UH of Nantes, Nantes
  - Hosptal of Saint Nazaire, Saint-Nazaire

REFERENCES:
- [Derived] Strullu M, Rakotonjanahary J, Tarral E, Savagner C, Thomas C, Mechinaud F, Reguerre Y, Poignant S, Boutet A, Bassil J, Medinger D, Quemener E, Young NL, Rachieru P, Klaassen RJ, Pellier I. Evaluation of health related quality of life in children with immune thrombocytopenia with the PedsQL 4.0 Generic Core Scales: a study on behalf of the pays de Loire pediatric hematology network. Health Qual Life Outcomes. 2013 Nov 13;11:193. doi: 10.1186/1477-7525-11-193. PMID 24225051